CLINICAL TRIAL: NCT06777004
Title: Predictive Factors of Analgesic Response in Patients With Pain Associated With Bone Metastasys: a Multicenter Prospective Observational Study
Brief Title: Predictive Factors of Analgesic Response in Patients With Pain Associated With Bone Metastasys
Acronym: CIBP
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CIBP
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Cancer Pain
Keywords: bone metastasis
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to improve the knowledge of pain associated with bone metastases, in particular to analyze the clinical course of patients who are affected by pain due to bone metastases, in order to better understand which factors may be related to a faster response to pain therapy.

DETAILED DESCRIPTION:
This is a non-profit, non-pharmacological, multicenter prospective observational study. Enrollment will last for 24 months from the opening of the study.

The overall duration of the study will be 36 months.

Based on the primary endpoint, patients will be stratified into 5 groups, corresponding to different times of achievement of stable pain:

1. patients who achieve stable pain at the first assessment (3 days)
2. patients who achieve stable pain at the second or third assessment (6-9 days)
3. patients who achieve stable pain at the fourth or fifth assessment (12-15 days)
4. patients who achieve stable pain at the sixth or seventh assessment (18-21 days)
5. patients who do not reach stable pain on the twenty-first day Based on the secondary endpoints, patients with and without neuropathic pain and with and without reaching PPG will be compared with the results of the HADS, EORT-QLQ-C30 [11] and Karnofsky scale [12-13] tests, in terms of final MEDD (morphine equivalent daily opioid dose) and type of drugs taken.

Enrolled patients will undergo validated tests, administered by appropriately trained personnel. All the tests mentioned here are in use in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Obtaining informed consent; age greater than or equal to 18 years definite diagnosis of solid tumor (histological and/or radiological, as indicated by the corresponding guidelines), already in charge of an Oncology service. bone metastases at any site, regardless of the type of primary tumor; patient with pain related to established, new-onset, or current bone metastases of the recrudescence of painful symptoms Enrollment must occur at the time of requesting medical intervention for pain related to bone lesions, within 72 hours of reporting.

Exclusion Criteria:

patients with cognitive and/or conscious impairments that could affect the evaluation; Patients with a history of substance/alcohol abuse/dependence or conditions that contraindicate administration of opioid analgesics; presence of non-oncological pathologies in the decompensation phase. non-understanding of the Italian language, both spoken and written.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who arrive within 24 months starting from February 2022 will be enrolled to the observation of one of the Centers participating in the study. A total population of about 200 patients is expected, a number based on an estimate retrospective on patients belonging to our Center.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Identify what are the possible factors associated with a faster achievement of stable pain. | From enrollment to 21 days following the start of analgesic treatment
  Specifically, the presence of a possible association between the analgesic response and factors related to the patient (clinical, demographic and laboratory), the neoplasm, the characteristics of symptomatic bone lesions and the results of the tests administered to the patient at enrollment and at the end-of-study visit will be sought.
  Primary end-point: addition of stable pain (NRS never greater than 3/10, for three consecutive days, with less than 3 intakes of analgesic therapy as needed (rescue dose) on each of these three days)

SECONDARY OUTCOMES:
To evaluate the incidence of neuropathic pain associated with bone metastases and its influence on the anxiety domain, quality of life, and patient autonomy. | From enrollment to 21 days following the start of analgesic treatment
  Incidence of neuropathic pain, defined based on the LANSS screening test and NeuPSIG guideline diagnostic algorithm.
  Whether or not PPG (personalized pain goal) is met

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lenzi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Irccs Azienda Ospedaliero Universitario Di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No